CLINICAL TRIAL: NCT06805578
Title: Exploring and Evaluating the Impact of 'Refresh and Reconnect!': A Museum-based Heritage Programme for Older Persons With Cognitive Impairment
Brief Title: Exploring and Evaluating the Impact of 'Refresh and Reconnect!'
Acronym: ReCognition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: National Heritage Board, Singapore (Unknown); National Museum Singapore, Singapore (Unknown)
Responsible Party: Principal Investigator, Rahul Malhotra, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2024-259
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Mild Cognitive Impairment (MCI); Ageing; Mild Dementia; Well-being
Keywords: Social Prescription; Heritage; Museum; Mild Cognitive Impairment; Mild Dementia; Person with cognitive impairment; Artist
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This is an exploratory study that adopts a quasi-experimental (single-arm, before-after) and mixed-methods quantitative and qualitative design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Persons with cognitive impairment will undergo a 6-week heritage-based intervention programme conducted by the National Museum of Singapore, which includes guided gallery tours led by the museum's Care Facilitator volunteers and artist-led hands-on activities based on various art forms.
  Interventions: Other: Heritage art programme

INTERVENTIONS:
Other: Heritage art programme — The 6-week 'Refresh and Reconnect!' programme includes guided gallery tours led by the museum's Care Facilitator volunteers and artist-led hands-on activities based on various art forms (e.g. artist-led dance, art, or drama workshops).
  Other Names: "Refresh and Reconnect!"

SUMMARY:
Dementia and mild cognitive impairment are a rising concern for the ageing population in Singapore, leading to diminished quality of life and health outcomes. Arts-based interventions in a museum setting have been shown to improve cognitive health and well-being for Persons with Cognitive Impairment (PWCIs), however little is known about the relationship of heritage-based interventions on the health and well-being of PWCIs.

This mixed-methods study evaluates the 6-week "Refresh and Reconnect!" programme (R&R!), a museum-based heritage programme including guided artist-led activities and tours of the National Museum of Singapore.

(i) In the quantitative study (n = 64-120 PWCIs, comprising with mild cognitive impairment (MCI) or mild dementia), assessments will be conducted at 2 time points (pre-programme, post-programme) to evaluate change in cognitive, social, and mental well-being.

ii) In the qualitative study, ethnographic observations of the R&R! programme; ethnographic interviews with staff (n= max 3), & artists (n= max 6); and in-depth interviews with PWCIs (n=16) will be used to elicit the underlying context-mechanisms-outcomes which enable R&R! success. Programme volunteers will also be engaged through casual or informal conversations as part of the ethnographic observations.

The study will provide valuable insights for the development of effective, non-pharmacological interventions for PWCIs. The primary objectives of the study are to (a) compare the change (before and after programme participation) in the health and well-being of PWCIs participating in the programme, and (b) assess the change (before and after programme participation) in the perception of the museum, 'heritage' and learning among PWCIs participating in the programme. The secondary aims are to understand the factors, contexts, and mechanisms that influence the implementation of the museum-based intervention and its effects, including the place-based effects of the curated museum Reunion space for PWCIs.

Achieving the objectives will help answer the following research questions:

1. To what extent, and how does participation in the "Refresh and Reconnect!" programme impact health and well-being of PWCIs?
2. To what extent, and how does participation in the programme affect the study participants' understanding and perception of the museum as a potential place to enhance one's health and well-being? [Note: Study Participants include all who are participating in the study such as PWCIs and those who are implementing (e.g. museum staff), facilitating (e.g. artists) and assisting (e.g. volunteers) with the R&R! Programme]
3. What are the contexts and mechanisms that influence the implementation of the programme?

These findings are of significant public health importance for Singapore, potentially informing policy decisions, resource allocation, and healthcare strategies to better support PWCIs, ultimately improving their quality of life. Findings of the study may also contribute to similar heritage-based programmes in future, contributing to the understanding of key elements of programme success, and for whom these programmes are effective for.

ELIGIBILITY:
Inclusion Criteria:

* Fulfils the programme recruitment criteria and registers for the programme through National Museum of Singapore's collaborating partners; AND
* Provides consent for participation in the study personally; AND
* Willing and able to participate in interviews independently, without proxy; AND
* Scores between 22 to 27 on the MoCA (or 22 to 26 for participants with less than 10 years of education; or 22 to 25 for participants who are unable to provide information on the number of years of formal education completed). These thresholds follow the recommendation of MoCA use in determining mild cognitive impairment and mild dementia in Singapore and draw from studies concerning mental capacity and consent for persons living with cognitive impairment

Exclusion Criteria:

* Whose cognitive impairment status cannot be confirmed by the administered screener; OR
* Do not give consent to participate in the study; OR
* Scores below 22 on the MoCA, or above 27 (or 26 for participants with less than 10 years of education; or 25 for participants who are unable to provide information on the number of years of formal education completed)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Quality of life at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Quality of life (QoL) will be assessed using the Control, Autonomy, Self-Realization, and Pleasure-11-SG (CASP-11-SG) scale. CASP-11-SG has been validated in Singapore. It has 11 items covering two domains: Control-Autonomy, and Self-realization-Pleasure (Table 1). Items are scored on a four-point response scale [Often (score = 3), Sometimes, Not Often, Never (score = 0)] based on how often the participant feels the way described in the item. Negatively worded items are reverse-coded. A higher total score (range: 0-33) indicates higher QoL. Control-Autonomy subscale (range: 0-18) and Self-realization-Pleasure subscale (range: 0-15) scores are also calculated.
Change from baseline in Health-related Quality of life at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Health-related Quality of life (HRQoL) will be assessed using the EuroQol- 5 Dimension (EQ-5D) questionnaire. The EQ-5D comprises five questions on mobility, self-care, pain, usual activities, and psychological status with five possible answers for each item (1=no problem, 2=slight problem, 3=moderate problem, 4=severe problem, 5=unable to do). Overall, a total score of 5 indicates the best health state, whereas higher scores indicate more severe or frequent problems. In addition, there is a visual analogue of the scale to indicate general health status, with a score of 100 indicating the best health status.
Change from baseline in anxiety and depression at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS). It is a self-reported rating scale of 14 items on a 4-point Likert scale (range 0-3), with 7 items each for anxiety and depression. The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Scores of 11 or more on either subscale are a significant 'case' of psychological morbidity, while scores of 8-10 represents 'borderline' and 0-7 'normal'.
Change from baseline in loneliness at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Loneliness will be assessed using The Three-Item Loneliness Scale. Each item of the scale has a five-point Likert response option: "Always" (scored as 4) "Fairly Often" (3), "Occasionally" (2), "Rarely" (1), and "Never" (scored as 0). The scores for each individual question can be added together to give a possible range of scores from 0 to 12. Higher scores indicate greater degrees of loneliness.
Change from baseline in social isolation at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Lubbens Social Network Scale 6-item (LSNS-6) is a social engagement scale that consists of six items. The score for each item ranges from 0 to 5, with 0 indicating none and 5 indicating nine or more. The total score is calculated by finding the sum of all items, and ranges from 0 to 30. A higher score indicates more social engagement.
Change from baseline in ageing perceptions at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  The Brief Ageing Perceptions Questionnaire (Brief-APQ) measure comprise Likert scale items that represent seven ageing perception domains. Participants rate their agreement with a series of statements - for example "I am always aware of my age" or "As I get older I can take part in fewer activities" with a five-point response scale with the options: Strongly Disagree, Disagree, Neither Agree nor Disagree, Agree, Strongly Agree.
Change from baseline in motivations to learn at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Motivations to learn will be assessed using the Readiness-to-learn Scale from the background questionnaire of the Programme for the International Assessment of Adult Competencies (PIAAC). This scale assesses participants' motivations to learn, and the learning strategies they adopt to solve challenges in learning. The response categories for this item range from not at all (1), to a very high extent (5).
Change from baseline in Montreal Cognitive Assessment score at the end of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Cognitive performance will be assessed using the Montreal Cognitive assessment (MoCA). MoCA assessment parameters are visuospatial/ executive, naming ability, vigilance, verbal fluency, delayed recall, and abstractions. The maximum MoCA score is 30 points. MCI (Mild Cognitive Impairment) is indicated by a score of less than 27 for those with 10 or more years of education or a score of less than 26 for those with less than 10 years of education (following the recommendation of MoCA use in Singapore).

SECONDARY OUTCOMES:
Changes to subjective well-being after each session of the 6-week intervention | From enrolment to the end of intervention at 6 weeks
  Museum-based subjective well-being will be assessed by University College London (UCL) Museum Wellbeing Measures toolkit. The toolkit includes a 12-item Generic Wellbeing Questionnaire (GWQ) and Positive Wellbeing Measures Umbrella, designed specifically for museum projects. The GWQ uses statements that refer to an emotion or life quality that participants might have experienced during the museum activity, such as 'I felt confident'. These are rated from 1 ('None of the time') to 5 ('All of the time'). The Positive Wellbeing Umbrella consist of a hexagonal shape with six sections of different colours. Each of the six sections has a word next to it related to a wellbeing mood or emotion and responses are ranged from one (I don't feel) to five (I feel extremely). Participants are required to rate the extent they feel the wellbeing word at that moment in time by circling the appropriate number.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Malhotra, MD, MPH, Principal Investigator — Duke-NUS Graduate Medical School; Ad Maulod, PhD, MSc, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- National Museum of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The investigator team will decide on sharing of individual participant data on a case-to-case basis, when such requests are made.

REFERENCES:
- [Background] Zietlow KE, Oyeyemi DM, Cook SE, Hardy M, McDonald SR, Lagoo-Deenadayalan S, Heflin MT, Whitson HE. RESEARCHCognition and Capacity to Consent for Elective Surgery. J Am Geriatr Soc. 2020 Nov;68(11):2694-2696. doi: 10.1111/jgs.16786. Epub 2020 Aug 17. No abstract available. PMID 33460037
- [Background] Yang M, Samper-Ternent R, Volpi E, Green AN, Lichtenstein M, Araujo K, Borek P, Charpentier P, Dziura J, Gill TM, Galloway R, Greene EJ, Lenoir K, Peduzzi P, Meng C, Reese J, Shelton A, Skokos EA, Summapund J, Unger E, Reuben DB, Williamson JD, Stevens AB. The dementia care study (D-CARE): Recruitment strategies and demographic characteristics of participants in a pragmatic randomized trial of dementia care. Alzheimers Dement. 2024 Apr;20(4):2575-2588. doi: 10.1002/alz.13698. Epub 2024 Feb 15. PMID 38358084
- [Background] Wu CY, Hung SJ, Lin KC, Chen KH, Chen P, Tsay PK. Responsiveness, Minimal Clinically Important Difference, and Validity of the MoCA in Stroke Rehabilitation. Occup Ther Int. 2019 Apr 14;2019:2517658. doi: 10.1155/2019/2517658. eCollection 2019. PMID 31097928
- [Background] Wu VX, Chi Y, Lee JK, Goh HS, Chen DYM, Haugan G, Chao FFT, Klainin-Yobas P. The effect of dance interventions on cognition, neuroplasticity, physical function, depression, and quality of life for older adults with mild cognitive impairment: A systematic review and meta-analysis. Int J Nurs Stud. 2021 Oct;122:104025. doi: 10.1016/j.ijnurstu.2021.104025. Epub 2021 Jun 30. PMID 34298320
- [Background] Veretennikoff K, Walker D, Biggs V, Robinson G. Changes in Cognition and Decision Making Capacity Following Brain Tumour Resection: Illustrated with Two Cases. Brain Sci. 2017 Sep 24;7(10):122. doi: 10.3390/brainsci7100122. PMID 28946652
- [Background] Teri L, Truax P, Logsdon R, Uomoto J, Zarit S, Vitaliano PP. Assessment of behavioral problems in dementia: the revised memory and behavior problems checklist. Psychol Aging. 1992 Dec;7(4):622-31. doi: 10.1037//0882-7974.7.4.622. PMID 1466831
- [Background] Tan SY, Lew KJ, Xie Y, Lee PSS, Koh HL, Ding YY, Lee ES. Healthcare cost of patients with multiple chronic diseases in Singapore public primary care setting. Ann Acad Med Singap. 2021 Nov;50(11):809-817. doi: 10.47102/annals-acadmedsg.2021246. PMID 34877584
- [Background] Tan LT, Ostbye T, Visaria A, Malhotra R. Derivation, and establishment of the validity and reliability, of the CASP-11-SG quality of life scale among community-dwelling older adults. Qual Life Res. 2023 Jan;32(1):295-306. doi: 10.1007/s11136-022-03238-4. Epub 2022 Sep 6. PMID 36068420
- [Background] Subramaniam M, Chong SA, Vaingankar JA, Abdin E, Chua BY, Chua HC, Eng GK, Heng D, Hia SB, Huang W, Jeyagurunathana A, Kua J, Lee SP, Mahendran R, Magadi H, Malladi S, McCrone P, Pang S, Picco L, Sagayadevan V, Sambasivam R, Seng KH, Seow E, Shafie S, Shahwan S, Tan LL, Yap M, Zhang Y, Ng LL, Prince M. Prevalence of Dementia in People Aged 60 Years and Above: Results from the WiSE Study. J Alzheimers Dis. 2015;45(4):1127-38. doi: 10.3233/JAD-142769. PMID 25672767
- [Background] Siow JYM, Chan A, Ostbye T, Cheng GH, Malhotra R. Validity and Reliability of the Positive Aspects of Caregiving (PAC) Scale and Development of Its Shorter Version (S-PAC) Among Family Caregivers of Older Adults. Gerontologist. 2017 Aug 1;57(4):e75-e84. doi: 10.1093/geront/gnw198. PMID 28082275
- [Background] Reschke-Hernandez AE, Gfeller K, Oleson J, Tranel D. Music Therapy Increases Social and Emotional Well-Being in Persons With Dementia: A Randomized Clinical Crossover Trial Comparing Singing to Verbal Discussion. J Music Ther. 2023 Oct 7;60(3):314-342. doi: 10.1093/jmt/thad015. PMID 37220880
- [Background] Poulos RG, Marwood S, Harkin D, Opher S, Clift S, Cole AMD, Rhee J, Beilharz K, Poulos CJ. Arts on prescription for community-dwelling older people with a range of health and wellness needs. Health Soc Care Community. 2019 Mar;27(2):483-492. doi: 10.1111/hsc.12669. Epub 2018 Oct 21. PMID 30345578
- [Background] Peters S, Lohse KR, Klassen TD, Liu-Ambrose T, Dukelow SP, Bayley MT, Hill MD, Pooyania S, Yao J, Eng JJ. Higher intensity walking improves global cognition during inpatient rehabilitation: a secondary analysis of a randomized control trial. Front Neurol. 2023 Jun 9;14:1023488. doi: 10.3389/fneur.2023.1023488. eCollection 2023. PMID 37360352
- [Background] Nowell, L. S., Norris, J. M., White, D. E., & Moules, N. J. (2017). Thematic Analysis: Striving to Meet the Trustworthiness Criteria. International Journal of Qualitative Methods, 16(1). https://doi.org/10.1177/1609406917733847
- [Background] Ng A, Chew I, Narasimhalu K, Kandiah N. Effectiveness of Montreal Cognitive Assessment for the diagnosis of mild cognitive impairment and mild Alzheimer's disease in Singapore. Singapore Med J. 2013 Nov;54(11):616-9. doi: 10.11622/smedj.2013220. PMID 24276096
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] National Population and Talent Division (2023). Population in Brief 2023: Key Trends. Strategy Group, Prime Minister's Office. https://www.population.gov.sg/media-centre/articles/population-in-brief-2023-key-trends/
- [Background] Musek, J., Polic, M. (2014). Personal Well-Being. In: Michalos, A.C. (eds) Encyclopaedia of Quality of Life and Well-Being Research. Springer, Dordrecht. https://doi.org/10.1007/978-94-007-0753-5_2148
- [Background] Mollers T, Perna L, Stocker H, Ihle P, Schubert I, Schottker B, Frolich L, Bauer J, Brenner H. Alzheimer's disease medication and outcomes of hospitalisation among patients with dementia. Epidemiol Psychiatr Sci. 2019 Nov 14;29:e73. doi: 10.1017/S2045796019000702. PMID 31722770
- [Background] Karlawish J, Cary M, Moelter ST, Siderowf A, Sullo E, Xie S, Weintraub D. Cognitive impairment and PD patients' capacity to consent to research. Neurology. 2013 Aug 27;81(9):801-7. doi: 10.1212/WNL.0b013e3182a05ba5. Epub 2013 Jul 26. PMID 23892706
- [Background] Jiao Y, Liu C, Chang J, Zhou S, Ji Y. Self-management preferences in patients with mild cognitive impairment: A qualitative study. Front Psychol. 2022 Oct 14;13:955960. doi: 10.3389/fpsyg.2022.955960. eCollection 2022. PMID 36312202
- [Background] Ito E, Nouchi R, Dinet J, Cheng CH, Husebo BS. The Effect of Music-Based Intervention on General Cognitive and Executive Functions, and Episodic Memory in People with Mild Cognitive Impairment and Dementia: A Systematic Review and Meta-Analysis of Recent Randomized Controlled Trials. Healthcare (Basel). 2022 Aug 3;10(8):1462. doi: 10.3390/healthcare10081462. PMID 36011119
- [Background] Hawkley LC, Browne MW, Cacioppo JT. How can I connect with thee? Let me count the ways. Psychol Sci. 2005 Oct;16(10):798-804. doi: 10.1111/j.1467-9280.2005.01617.x. PMID 16181443
- [Background] Gorges, J., Maehler, D.B., Koch, T., & Offerhaus, J. (2016). Who likes to learn new things: measuring adult motivation to learn with PIAAC data from 21 countries. Large-scale Assessments in Education, 4, 9. https://doi.org/10.1186/s40536-016-0024-4
- [Background] Gordon MF, Lenderking WR, Duhig A, Chandler J, Lundy JJ, Miller DS, Piault-Louis E, Doody RS, Galasko D, Gauthier S, Frank L; Patient-Reported Outcome Consortium's Cognition Working Group. Development of a patient-reported outcome instrument to assess complex activities of daily living and interpersonal functioning in persons with mild cognitive impairment: The qualitative research phase. Alzheimers Dement. 2016 Jan;12(1):75-84. doi: 10.1016/j.jalz.2015.04.008. Epub 2015 Jun 13. PMID 26079412
- [Background] Givon Schaham N, Buckman Z, Rand D. TECH preserves global cognition of older adults with MCI compared with a control group: a randomized controlled trial. Aging Clin Exp Res. 2024 Jan 20;36(1):1. doi: 10.1007/s40520-023-02659-6. PMID 38252189
- [Background] Forward Singapore Workgroup. (2023). Building our shared future. https://www.forwardsingapore.gov.sg
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Dinius CJ, Pocknell CE, Caffrey MP, Roche RAP. Cognitive interventions for memory and psychological well-being in aging and dementias. Front Psychol. 2023 Feb 2;14:1070012. doi: 10.3389/fpsyg.2023.1070012. eCollection 2023. PMID 36818134
- [Background] Cowan, B., Laird, R., & McKeown, J. (2019). Museum Objects, Health and Healing: The Relationship between Exhibitions and Wellness (1st ed.). Routledge. https://doi.org/10.4324/9780429467813
- [Background] Cobb, G.H. (2022). Understanding adult play and wellbeing in children's museums. MuseumsForward, 2(4).
- [Background] Chiang KJ, Chu H, Chang HJ, Chung MH, Chen CH, Chiou HY, Chou KR. The effects of reminiscence therapy on psychological well-being, depression, and loneliness among the institutionalized aged. Int J Geriatr Psychiatry. 2010 Apr;25(4):380-8. doi: 10.1002/gps.2350. PMID 19697299
- [Background] Bennington, R., Backos, A., Harrison, J., Etherington Reader, A., & Carolan, R. (2016). Art therapy in art museums: Promoting social connectedness and psychological well-being of older adults. The Arts in Psychotherapy, 49, 34-43. https://doi.org/10.1016/j.aip.2016.05.013
- [Background] An S, Ko J, Yu KS, Kwon H, Kim S, Hong J, Kong HJ. Exploring the Category and Use Cases on Digital Therapeutic Methodologies. Healthc Inform Res. 2023 Jul;29(3):190-198. doi: 10.4258/hir.2023.29.3.190. Epub 2023 Jul 31. PMID 37591674
- [Background] Baumann, J., Biscoe, N., Burnell, K., Lobban, J., & Murphy, D. (2023). Museum-based art therapy and wellbeing programme: experiences of veterans with PTSD1. International Journal of Art Therapy, 28(3), 142-149. https://doi.org/10.1080/17454832.2023.2188409

DOCUMENTS (2):
  • Study Protocol (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT06805578/Prot_000.pdf
  • Informed Consent Form (2025-01-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT06805578/ICF_001.pdf